CLINICAL TRIAL: NCT03982537
Title: Effect of N-Acetyl Cysteine (NAC) on the Oral Microbiome and on the Degree of Mucositis Developed in Response to Concurrent Chemotherapy and Radiotherapy in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Effect of N-Acetyl Cysteine (NAC) on the Oral Microbiome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Concept is withdrawn and a different concept will be submitted the near future.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00058729; WFBCCC 97119 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2019-06-05; First posted 2019-06-11 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck squamous cell cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Acetylcysteine; Drug Therapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nature's Blend N-Acetyl-L-Cysteine 600 mg with Chemotherapy (Experimental): The treatment with NAC will be given twice daily for at least 10 days with the goal to cover the window of opportunity time between the treatment decision for CRT and the beginning of treatment (usually 14-21 days).
  Interventions: Drug: N-Acetyl-L-Cysteine dietary supplement; Radiation: Chemotherapy and Radiation
- Standard of Care Chemotherapy (CONTROL) (Other): Patients will receive definitive or adjuvant concurrent chemotherapy and radiotherapy as per standard of care
  Interventions: Radiation: Chemotherapy and Radiation

INTERVENTIONS:
Drug: N-Acetyl-L-Cysteine dietary supplement — Treatment will be administered on an outpatient basis, either twice daily or 48 hours prior to starting chemotherapy radiation. Eligible participants will start NAC at least 9 days before definitive or adjuvant radiation therapy.
  Other Names: N-Acetyl-L-Cysteine
  Arms: Nature's Blend N-Acetyl-L-Cysteine 600 mg with Chemotherapy
Radiation: Chemotherapy and Radiation — Participants will receive definitive or adjuvant concurrent chemotherapy and radiotherapy s per standard of care.

SUMMARY:
This is a Phase II treatment, randomized 3:1 ratio, open label clinical trial to study the effect of short duration administration of N-acetyl cysteine on oral microbiome and on mucositis caused by concurrent chemotherapy and radiotherapy.

DETAILED DESCRIPTION:
Primary Objective(s) I. To determine whether short duration pre-treatment with N-acetyl cysteine reduces the rate of severe mucositis that develops during the standard concurrent chemoradiotherapy in patients with locally advanced Head and Neck Squamous Cell Cancer.

Secondary Objective(s) I. Identify the effect of N-acetyl cysteine on the oral microbiome.

II. Identify the effect of short duration pre-treatment with N-acetyl cysteine on the duration and delay onset of severe radiation-induced mucositis developed during the standard concurrent chemoradiotherapy in patients with locally advanced Head and Neck Squamous Cell Cancer.

III. Bank saliva and blood for future studies of biomarkers that will be correlated with changes in the oral microbiome and the duration of mucositis.

IV. Determine if there is any effect of short duration pre-treatment with N-acetyl cysteine on tumor response to standard CRT as measured within the first year of treatment.

V. Determine the relationship between human papillomavirus status and smoking status and the baseline microbiome as well as well as the possible differential effect of N-acetyl cysteine on the structure of the oral microbiome in human papillomavirus positive patients vs smokers.

VI. Gather data on the incidence, severity, duration and onset of severe radiation-induced mucositis as well as data on saliva and blood biomarkers and evaluation of the oral microbiome in patients receiving standard of care primary or adjuvant chemoradiotherapy to gather preliminary data for use in designing future Phase 3 studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed HNSCC.
* Patients must be scheduled for definitive or adjuvant concurrent drug therapy and radiotherapy to include the oral cavity in the field and have a window of at least 14 days between the treatment decision and beginning of treatment.
* Patients must be ≥ 18 years old.
* Willing to provide consent for collection of samples of blood and saliva as scheduled through the treatment.
* Subject is willing and able to comply with the protocol for the duration of the study.
* Ability to understand and the willingness to sign an IRB-approved informed consent document.

Exclusion Criteria:

* Patients who have used NAC as a supplement or as a treatment within the last 6 months.
* Patients who have participated in another clinical study with an investigational product during the last 8 weeks.
* Receipt of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) within the last 8 weeks.
* Patients who are unable to swallow pills.
* Patients Patient is on medications that need to be continued and that might interact with NAC.
* Uncontrolled pre-existent illness of the digestive tract such as PUD, GERD.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Reduction in Severe Mucositis with Pre-treatment N-acetyl cysteine | 3 months post treatment
  Severe mucositis will be defined as Grade III or IV mucositis as per WHO OM classification.

SECONDARY OUTCOMES:
Effects of N-acetyl cysteine on oral microbiome | At baseline and one year post treatment
  Oral microbiome profiling will be determined using 16S rRNA gene sequencing to characterize the bacterial diversity and composition in the saliva collected from participants before and after treatment.
Effects of standard of care chemoradiotherapy on oral microbiome | At baseline and one year post treatment
  Oral microbiome profiling will be determined using 16S rRNA gene sequencing to characterize the bacterial diversity and composition in the saliva collected from participants before and after treatment.
Number of Incidences of Severe Mucositis on N-acetyl cysteine | One year post treatment
  Time of development of mucositis grade III or above (marked as treatment day) and time of resolution below grade III (marked as post-treatment day) will be recorded and will serve to measure duration and delay onset of severe mucositis. For the time to event data, Kaplan Meier curves will be constructed to determine the median time to occurrence of severe mucositis.
Number of Incidences of Severe Mucositis with Standard of Care Chemoradiotherapy | One year post treatment
  Time of development of mucositis grade III or above (marked as treatment day) and time of resolution below grade III (marked as post-treatment day) will be recorded and will serve to measure duration and delay onset of severe mucositis
Number of Participants with Change in Saliva Biomarkers - N-acetyl cysteine | At baseline and one year post treatment
  Banked saliva to describe biomarkers that could correlate with oral microbiome changes and with the severity of mucositis. Measurements that would be considered are evaluations of the nitrate reducing and NO producing capacity of oral bacteria, saliva H2S measurements and metabolic profiling of saliva.
Number of Participants with Change in Saliva Biomarkers - Standard of Care Chemoradiotherapy | At baseline and one year post treatment
  Banked saliva to describe biomarkers that could correlate with oral microbiome changes and with the severity of mucositis. Measurements that would be considered are evaluations of the nitrate reducing and NO producing capacity of oral bacteria, saliva H2S measurements and metabolic profiling of saliva.
Number of Participants with Change in Blood Biomarkers - N-acetyl cysteine | At baseline and one year post treatment
  Blood samples to describe biomarkers that could correlate with oral microbiome changes and with the severity of mucositis. Measurements that would be considered are evaluations of the nitrate reducing and NO producing capacity of oral bacteria, saliva H2S measurements and metabolic profiling of blood.
Number of Participants with Change in Blood Biomarkers - Standard of Care Chemoradiotherapy | At baseline and one year post treatment
  Blood samples to describe biomarkers that could correlate with oral microbiome changes and with the severity of mucositis. Measurements that would be considered are evaluations of the nitrate reducing and NO producing capacity of oral bacteria, saliva H2S measurements and metabolic profiling of blood.
Tumor Response | One year post treatment
  Results of standard imaging studies and tumor response or progression will be collected from participant's electronic medical record and compared between participants pre-treated with N-acetyl cysteine and those no treated with N-acetyl cysteine.
Probability in Structure Changes of Microbiomes in Relation to Human Papillomavirus and Smoking Statuses and N-acetyl cysteine | One year post treatment
  Human papillomavirus status and smoking status at baseline will be examined and microbiome data collected over time will be compared between each group (i.e. smokers vs non-smokers) and (HPV+ vs HPV-) and then with both groups combined (smoker/HPV+, smoker/HPV-, non-smoker/HPV+ and non-smoker/HPV-) for continuous measures that describe the microbiome measures, a repeated measures mixed model will be used to make these comparisons where participants will be considered as random effects and HPV status, smoking status and time (and their interactions) will be considered as fixed effects.

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Porosnicu, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No